CLINICAL TRIAL: NCT00665249
Title: Component Analysis of Motivational Interviewing
Brief Title: Project Motion, A Study of Motivational Interviewing to Reduce Heavy or Problematic Drinking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Jonathan Morgenstern, Professor and Director, Substance Abuse Services, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R21AA017135-01 (NIH); R21AA017135-01 (NIH); NCT01117259 (obsolete NCT alias)
Record Dates: First submitted 2008-04-21; First posted 2008-04-23 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Alcohol Dependence; Alcohol Abuse
Keywords: problem drinking; heavy drinking; Alcohol; moderation; motivational interviewing
MeSH Terms: conditions — Alcoholism | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Full Motivational Interviewing (Active Comparator): This condition consisted of all the standard elements of MI, both the non-directive and directive strategies (Miller & Rollnick, 2002). Rogerian elements, such as warmth, egalitarianism, genuineness, and a client-centered approach to the therapeutic relationship, are commonly referred to as "MI Spirit" (Moyers, Martin, Manual, Hendricksen, & Miller, 2005). MI is comprised of MI spirit and includes specific directive strategies geared to focus the client toward targeted behavior change, such as confidence and importance rulers, visualization of behavior change, or a decisional balance. The directive elements of MI are those that selectively reinforce positive change talk or enhance discrepancy between a client's wish to change and stay with the status quo.
  Interventions: Behavioral: Motivational Interviewing
- No Intervention: Self Change (Active Comparator): Participants in this condition were not assigned to treatment, but were asked to attempt to change on their own during the 8-week follow-up period. SC participants were told that research had shown that some individuals could reduce their drinking without professional help; that participating in the IVR might facilitate their efforts; and that they would be offered professional treatment at the end of the 8-week period. As noted in the Introduction, SC was selected rather than a traditional wait-list control because the aim of the study was to decompose MI into its 3 hypothesized components that include self-change.
  Interventions: Other: Self-Change
- Spirit-Only Motivational Interviewing (Active Comparator): While this condition retained the Rogerian elements to MI, directive elements were excluded. For example, SOMI consisted of the non-directive elements including therapist stance (warmth, genuineness, egalitarianism), emphasis on client responsibility to change, extensive use of reflective listening skills (e.g., open-ended questions, simple reflections), and avoidance of MI-inconsistent behaviors (advise, confront, take expert role, interpretation). Reflective listening was focused on the whole experience of the client and the client's affect, and targeting a particular behavior or eliciting change talk about drinking was proscribed. Furthermore, tools utilized frequently in MI to develop discrepancy, such as amplified or double-sided reflections, were proscribed.
  Interventions: Behavioral: Spirit-Only Motivational Interviewing

INTERVENTIONS:
Behavioral: Motivational Interviewing — See MotivationalInterviewing.org
  Other Names: 4 one-hour Psychotherapy Sessions over 8 weeks.
  Arms: Full Motivational Interviewing
Behavioral: Spirit-Only Motivational Interviewing — Non-directive elements encompass the use of MI-consistent, and avoidance of MI-inconsistent, behaviors, as well as attention to MI-spirit.
  Other Names: SOMI; Non-Directive Psychotherapy
  Arms: Spirit-Only Motivational Interviewing
Other: Self-Change — Participants are followed for 8 weeks, without therapeutic intervention. At end of assessment period, they receive 4 sessions of full MI.
  Other Names: Waitlist Control
  Arms: No Intervention: Self Change

SUMMARY:
The purpose of this pilot study is to investigate the critical components of motivational interviewing (MI), a psychotherapeutic intervention, in reducing heavy or problematic drinking. The study will disaggregate MI into its component parts and test full MI compared to MI without its directive strategies. This study will test whether the directive elements of MI are critical or whether MI effects may be attributable solely to its Rogerian, non-directive components. For more information, go to www.projectmotion.org

DETAILED DESCRIPTION:
Motivational interviewing (MI) has been demonstrated to be an effective intervention for alcohol use disorders (AUD). The consistency, magnitude, and durability of its effects suggest powerful mechanisms of behavior change (MOBC) operate to reduce drinking. A better understanding of the MOBC in MI is therefore important. Existing MOBC studies of MI have yielded limited and contradictory findings. The project proposes to conduct a small pilot study to disaggregate MI into its component parts and test full MI compared to MI without its directive strategies. This test will compare whether the directive elements of MI (Full MI, or FMI) are critical or whether MI effects may be attributable solely to its Rogerian, non-directive components (aka, Spirit-Only MI, or SOMI).

In addition, we will test whether hypothesized main effects of FMI are mediated via increases in commitment to reduce drinking early in treatment. Further, we will examine whether non-specific therapy factors alone (SOMI) significantly reduce drinking when compared to a Feedback Followed by Counseling (FFC) condition that controls for non-therapy factors and incorporates assessment and self-monitoring. We will also test whether SOMI's main effects are mediated by increases in mood and greater belief in the ability to change, as hypothesized by various theories.

Our work on MOBC for MI will take place in the context of studying brief, stand-alone treatments for individuals with primary AUD who seek to reduce, but not stop, drinking. We will recruit 90 individuals with AUD seeking treatment; collect daily process data during a pre-treatment week; and then assess and randomly assign them to 3 conditions: FMI, SOMI, and FFC. All participants will be followed for 9 weeks using daily Interactive Voice Recording (IVR) and in-laboratory assessments at weeks 0, 1, 4, and 8. Those in treatment conditions will receive 4 sessions of treatment at weeks 1, 2, 4, and 8. FFC will receive treatment after completing the week 8 assessment period. Participants in FMI and SOMI will be followed for an additional 4 weeks post-treatment (week 12).

ELIGIBILITY:
Inclusion Criteria:

* age 18-65
* primary current diagnosis of alcohol use disorder
* have an average weekly consumption of >24 standard drinks (A standard drink is defined as 1.5 oz of 80 proof distilled spirits, a 5 oz. glass of wine, or a 12 oz. beer. These are all estimated to have about 0.5 oz or 9 grams of pure ethanol.)
* able to read English at the eighth grade or higher level and show no evidence of significant cognitive impairment
* are willing to reduce drinking to non-hazardous levels
* are willing to provide signed informed consent to participate
* agree not to seek additional substance abuse treatment during study period

Exclusion Criteria:

* have significant current substance use or substance dependence (with the exception of marijuana, nicotine and caffeine),defined as, any substance use (with the exception of marijuana, nicotine and caffeine) greater than weekly use in the past month
* have a serious psychiatric illness (e.g., psychotic disorder, bipolar disorder, major depression, etc.) or substantial suicide or violence risk
* having clinically severe alcoholism as evidenced by a history of significant medical problems associated with drinking, a history of seizures or severe withdrawal symptoms, or more than one inpatient treatment episode for drinking
* legally mandated to receive substance abuse treatment
* sufficiently socially unstable as to preclude completion of study requirements (e.g., homeless)
* state desire to pursue a goal of lifetime abstinence
* report current participation in or report an intent to participate in an additional substance abuse treatment method during the course of the study
* stated desire or intent to become pregnant or stated inconsistent use of birth control while sexually active

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2008-04; Primary Completion 2009-05 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Timeline Followback (TLFB)--Measures frequency and intensity of drinking by self-report | 8 weeks
  Daily record of drinking--measured in standard drink equivalents. The TLFB (Sobell, et al, 1980) assesses frequency of alcohol use during the previous 8 weeks. TLFB data is aggregated to provide weekly summary variables (sum of standard drinks per week, mean drinks per drinking day, and the mean number of drinking days) across the 8 weeks prior to randomization through the end of treatment. In order to compare baseline drinking, weekly summary variables were averaged across the 8 weeks prior to randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Jon Morgenstern, Ph.D., Principal Investigator — Columbia University; Alexis N Kuerbis, MSW, PhD, Study Director — Research Foundation for Mental Hygiene, Inc.
Locations (1):
- Research Foundation for Mental Hygiene, Inc., Columbia Addiction Services and Psychotherapy Intervention Research, New York, New York, United States

REFERENCES:
- See also: Project Motion — http://www.projectmotion.org